CLINICAL TRIAL: NCT04076306
Title: What is the Feasibility, Acceptability and Sensitivity of the iSTEP Exercise Test in Boys With Haemophilia?
Brief Title: What is the Feasibility of the ISTEP Exercise Test in Boys With Haemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16HI32
Record Dates: First submitted 2019-08-11; First posted 2019-09-03 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Accelerometry

STUDY DESIGN:
Intervention Model Description: Each child with haemophilia will undertake both the iSTEP exercise test and a modified shuttle walk test (10m-MSWT) in a randomised order on the same day with a washout period of at least 1 hour. This data will then be compared to previously collected normative data for the iSTEP test from healthy school age children from the original iSTEP development and validation study (Rand et al, 2015).
  The second component will include the feasibility of collecting standardised lower limb clinical muscle myometry measurements. The third component will be to explore the viability of collecting physical activity level data, in this population over a 7 day period using an accelerometer. This will be evaluated by monitoring the adherence to accelerometry wear. The value of the data will also be used to determine if it is useful at informing other aspects of fitness for boys with haemophilia.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iSTEP Feasibility Study Protocol (Other): All participants will be asked to undergo the entire protocol: iSTEP exercise test, 10 metre incremental shuttle walk test, myometry, accelerometry and Haemophilia Joint Health Score.
  Interventions: Other: iSTEP exercise testing

INTERVENTIONS:
Other: iSTEP exercise testing — iSTEP 10 minute step test, up and down on a commercial standard 3-height adjustable step Undertaking the 10m-MSWT 20-30 minutes Procedure takes place on testing track at Great Ormond Street Hospital; a 5 minute walk from the Haemophilia Centre. One of the research team accompanies the family with child to the track and will accompany them back to the Centre once testing is finished. Muscle Myometry 10 minutes, carried out by one of the research team at the end of the physiotherapy clinical assessment in the Haemophilia Centre. Wearing of accelerometer (activity/ step counter)7 days Device will be set up and provided at the end of the testing on the day of attendance at clinic. They will be instructed to wear this throughout the week at home when they are awake (at least 8 hours). Haemophilia Joint Health Score (HJHS) - a standardised outcome measure of joint health in people with Haemophilia, undertaken by the Clinical Specialist Physiotherapists in Haemophilia.
  Other Names: 10 metre Incremental Shuttle Walk Test; Muscle Myometry; Accelerometry; Haemophilia Joint Health Score (HJHS)

SUMMARY:
This study will be used to assess the feasibility and sensitivity of using the iSTEP, to assess exercise capacity in boys with haemophilia.

The feasibility criteria to be explored includes:

1. Recruitment to target number or better
2. The test procedure is completed within an allocated time (1-2 hours) and by 90% of participants without serious adverse events
3. 90% of participants achieve a sufficient exercise response (85% maximum heart rate (HRmax))
4. Calculation of estimates of minimum clinically important differences and variability for sample size calculations and responsiveness to severity of haemophilia and orthopaedic status The iSTEP exercise test will be compared to a more commonly used exercise test the modified shuttle walk test (10m- MSWT). Muscle strength (using myometry) will also be tested and compared to exercise performance for any relationships. Physical activity levels will also be assessed to obtain some baseline measurements of physical activity levels in this patient population, which are currently not very well known. The overarching aim of this current study is also to establish a robust and sensitive exercise test and to gain an understanding of the effects of physical activity levels and muscle strength on exercise capacity in this population.

DETAILED DESCRIPTION:
Identification of potential participants Eligible participants will be identified from the clinical patient database in the Haemophilia Centre at Great Ormond Street Hospital (GOSH) for Children NHS Trust. Potential participants will then be randomly selected. A simple randomisation approach will be employed using a computer random number table to select potential participants from the database. The parents / legal guardians will then be approached initially by the investigator via telephone to provide a brief verbal explanation of the research study and ask if they would be happy to receive a patient information sheet prior to their next clinic appointment. Should they be interested in participating in the study they will receive, by post, the PIS (one for parents and a separate age appropriate version for children) at least one week prior to their next clinic appointment. This will allow for a 'cooling-off' period of a minimum of one week for the potential participants. The researcher will then be available for questions by telephone or at the participant's next clinic appointment.

For the normal healthy control exercise test comparison population, data will be obtained from the existing iSTEP healthy control data collected as part of the iSTEP study from children in primary schools in London. This sample of 30 participants will be matched to the haemophilia group in terms of sex, age, body mass and stature.

Participant Recruitment

Consent of participants:

Most study recruits will be unable to give consent to participate due to their age. If the family have indicated that they are interested in participating in the study then at an agreed time (likely the next clinic appointment) one of the investigators from the research team will meet with the child participant and parent / legal guardian to complete the consent and assent forms as appropriate. The investigator will further explain the study procedures to the parent and child, why they are being asked to consider to be a part of the study and the associated risks and benefits of being included. The parent and child will then be given an opportunity to ask any further questions. The child/parent/legal guardian will then be asked to confirm if they agree to take part in the study. If consent is agreed a parental consent form will be completed by the parent/guardian and a copy will be provided. If the child assents then they will be asked to sign an assent form. If at any point during the study process the parent/guardian does not consent to inclusion in the study or the child withdraws their assent, then any data collected will be destroyed. Any decision to refuse or withdraw from the study will in no way influence the services that they receive.

Discussion with parents about the project will be undertaken with the child present. Once the child's parent/guardian has given consent, the child must also indicate that they do not object to participating in the research activity and understand what is involved. This participant 'assent' will be sought from participants in concordance with the legal requirements in England as set out in the following documents:

* Children Act 1989
* Medical Research Council (2004). MRC Ethics Guide: Medical research involving children. Version 3.2 May 2007 A signed participant assent form will be completed and a copy will be provided (Appendix 3).

The participant's medical team will be informed that they have volunteered to participate in this study, through verbal handover and documentation within the medical notes. Non-clinical members of the research team will only be able to access the participant's medical records once signed consent of this specific item has been provided.

The evaluation of the recruitment process will include recording of percentages of refusals to consent and stated reasons, as part of the feasibility aspect of this study. This will inform the design of future studies with this group with regards to approach and recruitment protocols. Confidentiality Data collection and storage will be undertaken in accordance with; The Caldicott Principles, Data Protection Act 1998 and Confidentiality: NHS Code of Practice 2003. The non-clinical members of the research team will only access data once consent has been provided from the parent/s. To ensure participant's confidentiality, data will be made anonymous by allocating a study participant number to identify their data. The research team will be the only ones to know the identity of each individual against his or her study number. All data will be recorded on a GOSH Trust computer under an electronic folder with restricted access for the investigators involved in the trial, electronic files will be encrypted and password protected. During the phases of data collection and analysis, only the chief investigator and research team will have access to the raw data and research findings. On completion of the research, data will be summarised and de-identified findings will be disseminated through publication in an appropriate professional journal and/or conference presentation.

Should a participant experience exacerbation to any joint pain during the exercise trial process, they will be able to stop and rest at any time. Should they feel unable to continue they will be able to withdraw from the study. The iSTEP is an exercise test that uses a step, which is tailored to the participant's height. It becomes incrementally more difficult every 2 minutes over the 10 minutes of the test, as the participant has to step up and down in time with a metronome (on audio track). The test ends when the participant is too tired to continue (see iSTEP protocol below), falls out of time with the metronome for stepping or at the end of the 10 minutes (that includes all 5 levels). Heart rate is taken at rest (before test), immediately afterwards and 3 minutes after the test.

The 10m- Modified Shuttle Walk Test (10m-MSWT) is a fitness bleep test that is also incremental. There are 25 levels, each level lasts 1 minute. The audio track guides the test, the bleeps at the beginning of the test are spaced widely apart (e.g. 20seconds to walk 10m in the first level). The time between bleeps becomes shorter every minute so that the participant will have to start fast walking then jogging at approximately level 6. At level 10 onwards the participant will need to run to keep in time with the bleeps. The test finishes when the participant is unable to continue due to , fatigue, breathlessness, or is unable to keep up with the bleeps. Heart rate is taken at rest, immediately after the test and 3 minutes after the test is finished (protocol below). Muscle myometry: uses a device to measure muscle power and is commonly used in research. The participant will be asked to push against resistance as strongly as they are able and the maximal power is calculated by the device (protocol below). Accelerometry: Activity will be measured using the ActiGraph GT3X, an accelerometer that measures volumes and patterns of activity. The ActiGraph has been extensively validated in children. A 15-second sampling epoch will be selected in order to optimize the ability to capture the sporadic nature of children's activity. Children will be asked to wear the accelerometer on an belt on the right hip for seven consecutive days during all waking hours. Accelerometers will be provided to families on the testing day and they will be asked to return it as soon as possible after the monitoring period (7days) using a supplied pre-paid envelope.

PROTOCOLS:

iSTEP Protocol Preparation

* The explanation to the participant is located on the pre-recorded audio track
* They will be required to step up and down in time with a metronome.

  - The height of the step is standardised for each child and will be based on approximately 50% of the length of the child's fibula.
* There is a bell to start. Thereafter the audio-track emits a metronome bleep at set speeds for 2 minutes at regularly spaced intervals.
* After every 2 minutes, the speed of stepping is increased by a small increment, so the participant steps progressively faster; the change in incremental stepping speed is indicated by a bell bleep.
* The first speed of walking is referred to as LEVEL 1, the second as LEVEL 2, and so on. Each level lasts for 2 minutes and the audio-recording continues for 5-levels (10 minutes in total). Each level contains a number of steps the number of which is dictated by the speed of that level.
* The first level reciprocally stepping up and down at a rate of 36
* To help the participant establish the first very slow speed of stepping, the operator steps alongside for the first time.

  4. End point of the test
* If the participant completes the 10 minutes (5 levels of the test) the test is completed.
* The end point of the test may be determined by the operator when:

  * Inability to maintain rhythm with the metronome, progressive speeding up and slowing down for >30 seconds
  * Loss of coordination
  * Light headedness
  * Extreme exhaustion
  * Sudden pallor
  * Undue signs of distress including severe wheezing or chest pain 10M MODIFIED SHUTTLE WALK TEST (25 LEVELS) PROTOCOL GENERAL INSTRUCTIONS Similar guidance to participants as provided for iSTEP Starting the test
* There is a triple bleep to start. Thereafter the audio-track emits a single bleep at regularly spaced intervals. The participant should aim to be at the opposite end to the start by the time the bleep sounds.
* After first minute, the speed of walking is increased by a small increment, so the participant walks progressively faster; the change in incremental speed is indicated by a triple bleep.
* The first speed of walking is referred to as LEVEL 1, the second as LEVEL 2, and so on. Each level lasts for 1 minute and the audio-recording continues for 25-levels. Each level contains a number of shuttles (10m in length), the number of which is dictated by the speed of that level. End point of the test
* The end point of the test may be determined by the participant:

When he or she becomes too breathless to maintain the required speed

• The end point of the test may be determined by the operator when: Undue signs of distress including severe wheezing or chest pain Failure of the patient to complete the shuttle in the time allowed. This test takes approximately 10-15 minutes, dependant on participant. MUSCLE MYOMETRY PROTOCOL A hand held dynamometer will be used to record the force produced by a maximum voluntary isometric contraction (MVIC) of the knee extensors, and ankle dorsi and plantar flexors. This test will take 5-10 minutes as part of their routine clinical examination. The total time required of the participant, on top of the routine clinic visit will be approximately 1 hour 30 minutes.

A14-1. In which aspects of the research process have you actively involved, or will you involve, patients, service users, and/or their carers, or members of the public? Design of the research Management of the research Undertaking the research Analysis of results Dissemination of findings None of the above Give details of involvement, or if none please justify the absence of involvement.

Parents and children were approached to provide comments and changes to the PIS forms in wording and design. In addition they provided opinion upon the potential burden of the of undertaking the testing. They reported that they did not feel the testing protocol sounded too onerous on top of normal clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Boys with mild, moderate and severe haemophilia aged 6 - 15 years (haemophilia A or B)
* Inhibitor or non-inhibitor
* Child able to follow simple verbal instructions, provide informed consent or assent

Exclusion Criteria:

* Child has a past history of acquired brain injury
* Child has a past history of any other disturbance of the central nervous system
* Joint or muscle bleed in the lower limb in the past 6 weeks
* Presence of lower limb pain on day of testing
* Diagnosis of severe asthma or exercise induced bronchoconstriction

Ages: 6 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of the study protocol, as measured by recruitment success. | 10 months
  Percentage of participants recruited from the number of approached.
Safety and Acceptability of the study protocol, as measured by the occurrence of any serious adverse events or reactions. | 10 months
  Evaluate whether the test procedure is completed within the allocated time (1-2 hours) without serious adverse events in >90% of participants.

SECONDARY OUTCOMES:
Pain before, during, immediately post and 3 mins post exercise tests | 5 minutes
  Subjective pain report; the Wong-Baker FACES Pain Rating Scale using a choice of 3 ways for the participant to report pain: Numerically; 0-10, 0 being no pain and 10 being the highest pain score; Pictorially, using faces representing level of pain; and words to describe lowest to highest pain levels eg: 'no hurt' to 'hurts worst'.
Time spent in moderate to vigorous activity | 7 days
  Accelerometry data
Muscle Myometry | 15 minutes.
  Using a hand-held dynamometer, a measure of the strength (in newton-metres, nm) of 3 different lower limb muscle groups; knee extensors, ankle plantarflexors and dorsiflexors.
Haemophilia Joint Health Score (HJHS) 2.1 | 30 minutes.
  A standardised measure of joint health used in routine assessment of children, young people and adults with Haemophilia, assessing 6 different joints, and gait, producing a score of 0-124. Lower scores indicate better joint health.
Duration exercise test completed in. | Typically, up to 15 minutes.
  For how long was the participant able to exercise, on the specified exercise test?

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Thorpe, Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Research and Development Office, Division of Research and Innovation,, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data made available to other researchers or statisticians for analysis.

REFERENCES:
- [Derived] Thorpe N, Harniess P, Main E, Hubert N, Rand S, Stephensen D, Liesner R, Bladen M. Feasibility, safety and acceptability of select outcome measures in a physiotherapy study protocol for boys with haemophilia. Pilot Feasibility Stud. 2021 May 6;7(1):105. doi: 10.1186/s40814-021-00831-1. PMID 33957997